CLINICAL TRIAL: NCT04612140
Title: STereotactic Ablative Radiosurgery of Recurrent Ventricular Tachycardia in Structural Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Institute for Clinical and Experimental Medicine (Other Government); Hospital Podlesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR-VT 2020
Record Dates: First submitted 2020-10-05; First posted 2020-11-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Ventricular Tachycardia
Keywords: Structural Heart Disease; Ventricular Tachycardia; Substrate Ablation; Stereotactic Radiosurgery; Functional Radiosurgery; 4D navigation
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomized into one of the two study arms.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiosurgery (Experimental): Eligible patients will be assigned to 2 treatment arms - radiosurgery (active arm) or repeated catheter ablation (control arm) in 1:1 fashion by covariate-adaptive randomization algorithm considering age, gender, etiology of SHD, LV ejection fraction, and serum NT-proBNP level.
  Interventions: Procedure: Radiosurgery
- Repeated catheter ablation (Active Comparator): Eligible patients will be assigned to 2 treatment arms - radiosurgery (active arm) or repeated catheter ablation (control arm) in 1:1 fashion by covariate-adaptive randomization algorithm considering age, gender, etiology of SHD, LV ejection fraction, and serum NT-proBNP level.
  Interventions: Procedure: Repeated catheter ablation

INTERVENTIONS:
Procedure: Radiosurgery — The study subjects randomized in this study arm will undergo a radiosurgery procedure.
  Arms: Radiosurgery
Procedure: Repeated catheter ablation — The study subjects randomized in this study arm will undergo repeated catheter ablation.
  Arms: Repeated catheter ablation

SUMMARY:
A multicentre trial on clinical effects of radiosurgical ablation of ventricular tachycardia (VT).

DETAILED DESCRIPTION:
Patients with previously failed conventional RF catheter ablation will be randomized to radiosurgery (active treatment group) or repeated catheter ablation (control treatment group). Details on inclusion and exclusion criteria are provided below.

Randomization Eligible patients will be assigned to 2 treatment arms - radiosurgery (active arm) or repeated catheter ablation (control arm) in 1:1 fashion by covariate-adaptive randomization algorithm considering age, gender, etiology of structural heart disease (SHD), left ventricular (LV) ejection fraction, and serum B-type natriuretic peptide (NT-proBNP) level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with structural heart disease (SHD) of any etiology (ischemic, non-ischemic, congenital corrected or uncorrected)
2. Implanted implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy-defibrillator (CRT-D)
3. Prior ≥1 catheter ablation procedure for VT due to SHD of them the last one performed in the expert center and employed:

   3.1 all meaningful mapping/ablation approaches (endocardial/epicardial access to left / right ventricular substrate as possible or appropriate) 3.2 precise electroanatomical mapping of the arrhythmogenic substrate in anticipation of future radiosurgery 3.3 additional mapping of structures used for precise image integration (aortic arch, left main ostium, right ventricular endocardial surface)
4. VT recurrence after the last catheter ablation fulfilling all criteria as follows:

   4.1 clinically relevant and requiring further intervention 4.2 compatible with the previously characterized arrhythmogenic substrate 4.3 occurred on stable antiarrhythmic medication (mostly amiodarone) unless contraindicated 4.4 reversible cause excluded
5. Signed an Institutional Review Board (IRB)-approved written informed consent

Exclusion Criteria:

1. Age < 20 years
2. Acute coronary syndrome or recent percutaneous coronary intervention or cardiac surgery (< 3 months)
3. Primary electrical disease (channelopathy)
4. Pregnancy or breastfeeding
5. Chronic heart failure with New York Heart Association (NYHA) Class IV
6. Serious comorbidities with presumed life expectancy less than one year
7. Significant peripheral artery disease precluding retrograde aortic mapping

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Recurrence of sustained VT after 3-month blanking period | 3 months
  Recurrence of sustained VT after 3-month blanking period will be assessed.

SECONDARY OUTCOMES:
VT burden according to implantable device | 3 months
  Number of sustained VT burden in three 3-month intervals after radiosurgery will be assessed.
Non-inducibility of VT at 6 months | 6 months
  TRUE/FALSE - Pacing protocol will be using 2 basic cycle length drives (600 and 400 ms) and 1-3 extrastimuli with coupling intervals decremented by 10 ms up to the refractoriness or 200 ms.
Recurrence of sustained VT excluding antitachycardia-pacing (ATP)-treated episodes | 24 months
  Recurrence of sustained VT excluding ATP-treated episodes will be assessed.
Electric storm recurrence | 24 months
  The recurrence of electric storm will be observed.
Cardiovascular hospitalization | 24 months
  The number of hospitalisations due to cardiovascular indications will be observed.
All-cause death | 24 months
  The all-cause death will be observed.
Change in quality of life: EQ-5D | 24 months
  Change in quality of life will be observed using the standardised EQ-5D (5-dimension) questionnaire. EQ-5D is a standardised instrument in the form of a questionnaire developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The quality of life is assessed in five dimensions, with three levels in each dimension. The higher score the patient achieves, the better the quality of life.
Change in echocardiographic indices | 24 months
  Left vetricle ejection fraction (%) will be observed.
Rate of major procedure-related complications (control arm) | 24 months
  The rate of major procedure-related complications will be observed among the study subjects enrolled to the control arm of the study, according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Rate of acute post-radiation complications (intervention arm) | 24 months
  The rate of acute post-radiation complications will be observed among the study subjects enrolled to the intervention arm of the study, according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)
Extent of scar | 6 months
  The extent of scar will be assessed 6 months after radiosurgery, based on invasive electroanatomical mapping.
Rate of late radiation-induced events | 24 months
  The rate of late radiation-induced events will be assessed according to CTCAE 5.0 in each cohort of isodose line level, specifically, rate of radiation myocarditis, pericarditis, and pneumonitis.
Radiation dose | 24 months
  The radiation dose will be observed for each interventional procedure, CT imaging and radiosurgery, together with the cumulative dose.
Need of antiemetic drugs | 24 months
  The need of antiemetic drugs will be assessed in all study subjects.
Dynamics of serum troponin level | 24 months
  The dynamics of serum troponin level will be observed in all study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Cvek, Ass.Prof.,MD,Ing, PhD,MBA, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - Hospital Podlesí, Třinec, Moravian-Silesian Region
  - Institute for Clinical and Experimental Medicine, Prague

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers, these may be made available upon request.

REFERENCES:
- [Background] Connolly SJ, Hallstrom AP, Cappato R, Schron EB, Kuck KH, Zipes DP, Greene HL, Boczor S, Domanski M, Follmann D, Gent M, Roberts RS. Meta-analysis of the implantable cardioverter defibrillator secondary prevention trials. AVID, CASH and CIDS studies. Antiarrhythmics vs Implantable Defibrillator study. Cardiac Arrest Study Hamburg . Canadian Implantable Defibrillator Study. Eur Heart J. 2000 Dec;21(24):2071-8. doi: 10.1053/euhj.2000.2476. PMID 11102258
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Connolly SJ, Dorian P, Roberts RS, Gent M, Bailin S, Fain ES, Thorpe K, Champagne J, Talajic M, Coutu B, Gronefeld GC, Hohnloser SH; Optimal Pharmacological Therapy in Cardioverter Defibrillator Patients (OPTIC) Investigators. Comparison of beta-blockers, amiodarone plus beta-blockers, or sotalol for prevention of shocks from implantable cardioverter defibrillators: the OPTIC Study: a randomized trial. JAMA. 2006 Jan 11;295(2):165-71. doi: 10.1001/jama.295.2.165. PMID 16403928
- [Background] Moss AJ, Schuger C, Beck CA, Brown MW, Cannom DS, Daubert JP, Estes NA 3rd, Greenberg H, Hall WJ, Huang DT, Kautzner J, Klein H, McNitt S, Olshansky B, Shoda M, Wilber D, Zareba W; MADIT-RIT Trial Investigators. Reduction in inappropriate therapy and mortality through ICD programming. N Engl J Med. 2012 Dec 13;367(24):2275-83. doi: 10.1056/NEJMoa1211107. Epub 2012 Nov 6. PMID 23131066
- [Background] Mallidi J, Nadkarni GN, Berger RD, Calkins H, Nazarian S. Meta-analysis of catheter ablation as an adjunct to medical therapy for treatment of ventricular tachycardia in patients with structural heart disease. Heart Rhythm. 2011 Apr;8(4):503-10. doi: 10.1016/j.hrthm.2010.12.015. Epub 2010 Dec 13. PMID 21147263
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Background] Aldhoon B, Wichterle D, Peichl P, Cihak R, Kautzner J. Outcomes of ventricular tachycardia ablation in patients with structural heart disease: The impact of electrical storm. PLoS One. 2017 Feb 10;12(2):e0171830. doi: 10.1371/journal.pone.0171830. eCollection 2017. PMID 28187168
- [Background] Raymond JM, Sacher F, Winslow R, Tedrow U, Stevenson WG. Catheter ablation for scar-related ventricular tachycardias. Curr Probl Cardiol. 2009 May;34(5):225-70. doi: 10.1016/j.cpcardiol.2009.01.002. PMID 19348944
- [Background] Kumar S, Baldinger SH, Romero J, Fujii A, Mahida SN, Tedrow UB, Stevenson WG. Substrate-Based Ablation Versus Ablation Guided by Activation and Entrainment Mapping for Ventricular Tachycardia: A Systematic Review and Meta-Analysis. J Cardiovasc Electrophysiol. 2016 Dec;27(12):1437-1447. doi: 10.1111/jce.13088. Epub 2016 Oct 6. PMID 27574120
- [Background] Jais P, Maury P, Khairy P, Sacher F, Nault I, Komatsu Y, Hocini M, Forclaz A, Jadidi AS, Weerasooryia R, Shah A, Derval N, Cochet H, Knecht S, Miyazaki S, Linton N, Rivard L, Wright M, Wilton SB, Scherr D, Pascale P, Roten L, Pederson M, Bordachar P, Laurent F, Kim SJ, Ritter P, Clementy J, Haissaguerre M. Elimination of local abnormal ventricular activities: a new end point for substrate modification in patients with scar-related ventricular tachycardia. Circulation. 2012 May 8;125(18):2184-96. doi: 10.1161/CIRCULATIONAHA.111.043216. Epub 2012 Apr 4. PMID 22492578
- [Background] Di Biase L, Santangeli P, Burkhardt DJ, Bai R, Mohanty P, Carbucicchio C, Dello Russo A, Casella M, Mohanty S, Pump A, Hongo R, Beheiry S, Pelargonio G, Santarelli P, Zucchetti M, Horton R, Sanchez JE, Elayi CS, Lakkireddy D, Tondo C, Natale A. Endo-epicardial homogenization of the scar versus limited substrate ablation for the treatment of electrical storms in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2012 Jul 10;60(2):132-41. doi: 10.1016/j.jacc.2012.03.044. PMID 22766340
- [Background] Tzou WS, Frankel DS, Hegeman T, Supple GE, Garcia FC, Santangeli P, Katz DF, Sauer WH, Marchlinski FE. Core isolation of critical arrhythmia elements for treatment of multiple scar-based ventricular tachycardias. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):353-61. doi: 10.1161/CIRCEP.114.002310. Epub 2015 Feb 13. PMID 25681389
- [Background] Tung R, Michowitz Y, Yu R, Mathuria N, Vaseghi M, Buch E, Bradfield J, Fujimura O, Gima J, Discepolo W, Mandapati R, Shivkumar K. Epicardial ablation of ventricular tachycardia: an institutional experience of safety and efficacy. Heart Rhythm. 2013 Apr;10(4):490-8. doi: 10.1016/j.hrthm.2012.12.013. Epub 2012 Dec 11. PMID 23246598
- [Background] Tokuda M, Kojodjojo P, Tung S, Tedrow UB, Nof E, Inada K, Koplan BA, Michaud GF, John RM, Epstein LM, Stevenson WG. Acute failure of catheter ablation for ventricular tachycardia due to structural heart disease: causes and significance. J Am Heart Assoc. 2013 May 31;2(3):e000072. doi: 10.1161/JAHA.113.000072. PMID 23727700
- [Background] Loo BW Jr, Soltys SG, Wang L, Lo A, Fahimian BP, Iagaru A, Norton L, Shan X, Gardner E, Fogarty T, Maguire P, Al-Ahmad A, Zei P. Stereotactic ablative radiotherapy for the treatment of refractory cardiac ventricular arrhythmia. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):748-50. doi: 10.1161/CIRCEP.115.002765. No abstract available. PMID 26082532
- [Background] Cuculich PS, Schill MR, Kashani R, Mutic S, Lang A, Cooper D, Faddis M, Gleva M, Noheria A, Smith TW, Hallahan D, Rudy Y, Robinson CG. Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia. N Engl J Med. 2017 Dec 14;377(24):2325-2336. doi: 10.1056/NEJMoa1613773. PMID 29236642
- [Background] Robinson CG, Samson PP, Moore KMS, Hugo GD, Knutson N, Mutic S, Goddu SM, Lang A, Cooper DH, Faddis M, Noheria A, Smith TW, Woodard PK, Gropler RJ, Hallahan DE, Rudy Y, Cuculich PS. Phase I/II Trial of Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia. Circulation. 2019 Jan 15;139(3):313-321. doi: 10.1161/CIRCULATIONAHA.118.038261. PMID 30586734
- [Background] Jumeau R, Ozsahin M, Schwitter J, Vallet V, Duclos F, Zeverino M, Moeckli R, Pruvot E, Bourhis J. Rescue procedure for an electrical storm using robotic non-invasive cardiac radio-ablation. Radiother Oncol. 2018 Aug;128(2):189-191. doi: 10.1016/j.radonc.2018.04.025. Epub 2018 May 9. PMID 29753550
- [Background] Haskova J, Peichl P, Pirk J, Cvek J, Neuwirth R, Kautzner J. Stereotactic radiosurgery as a treatment for recurrent ventricular tachycardia associated with cardiac fibroma. HeartRhythm Case Rep. 2018 Oct 24;5(1):44-47. doi: 10.1016/j.hrcr.2018.10.007. eCollection 2019 Jan. No abstract available. PMID 30693205
- [Background] Neuwirth R, Cvek J, Knybel L, Jiravsky O, Molenda L, Kodaj M, Fiala M, Peichl P, Feltl D, Januska J, Hecko J, Kautzner J. Stereotactic radiosurgery for ablation of ventricular tachycardia. Europace. 2019 Jul 1;21(7):1088-1095. doi: 10.1093/europace/euz133. PMID 31121018